CLINICAL TRIAL: NCT03456505
Title: Dissecting De-automatization: The Effect of Mindfulness Training on Unconscious Habit Formation
Brief Title: Dissecting De-automatization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Adam Hanley, Principal Investigator, University of Utah
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB_00088540
Record Dates: First submitted 2018-01-12; First posted 2018-03-07 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Mindfulness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): Participants randomly assigned to the mindfulness meditation condition will meet for five, 15-minute sessions, in which they will receive training in basic mindfulness skills (Wallace, 2006).
  Interventions: Behavioral: Mindfulness Meditation Training
- Active Listening (Active Comparator): Participants randomly assigned to the active listening condition will meet for five, 15-minute sessions, in which they will listen to Gilbert White's The Natural History of Selborne.
  Interventions: Behavioral: Active Listening

INTERVENTIONS:
Behavioral: Mindfulness Meditation Training — A researcher will guide participants through 5 mindfulness meditations, each lasting 11 minutes in length.
  Arms: Mindfulness
Behavioral: Active Listening — A researcher will read participants 5 selections from The Natural History of Selborne, each lasting 11 minutes in length.
  Arms: Active Listening

SUMMARY:
The proposed study will assess the effects of mindfulness meditation training on an eye blink conditioning (EBC) task in a sample of novice meditators. This methodology will allow investigation of whether mindfulness interrupts classical conditioning through the process of de-automatization. Implicit learning rates, as reflective of unconscious habit formation and measured by the frequency of conditioned responses during the EBC, will be a main outcome of interest. The proposed study will also assess the effects of mindfulness meditation training on an emotion regulation (ER) task, with a specific focus on reappraisal of negative images and savoring of positive images.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60,
2. willingness to participate in study interventions and assessments.

Exclusion Criteria:

1. Prior experience with Mindfulness-Based Stress Reduction, Mindfulness-Based Cognitive Therapy, or Mindfulness-Based Relapse Prevention, or a history of meditation practice,
2. Learning disability, significant memory problems or significant attentional disruptions as determined by self-report,
3. History of head injury resulting in loss of consciousness.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Conditioned Eyeblink Frequency | 9 minutes
  Between group differences in the frequency of conditioned eyeblinks over the six reinforcement blocks.

SECONDARY OUTCOMES:
Positive Emotion Regulation Task | 5 minutes
  Between group differences in affective change occasioned by savoring positive images will be measured by comparing increases in self-reported positive affect (5-point Likert scale) from pre- to post- positive image, viewing block.
Negative Emotion Regulation Task | 5 minutes
  Between group differences in affective change occasioned by positively reappraising negative images will be measured by comparing increases in self-reported negative affect (5-point Likert scale) from pre- to post- negative image, viewing block.
Self-Transcendence (NADA-State) | 2 minutes
  Between group differences in the degree to which mindfulness training alters participants' sense of self as measured by the nondaul awareness dimension assessment's (NADA) state form.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No